CLINICAL TRIAL: NCT05142293
Title: One Day Implantation Program for Heart Failure Patients Implanted With BIOTRONIK Cardiac Resynchronization Therapy Pacemakers
Brief Title: One Day Implantation Program for Heart Failure Patients Implanted With CRT-P
Acronym: OEDIPE-CRT-P
Status: Active, not recruiting | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR027
Record Dates: First submitted 2021-10-25; First posted 2021-12-02 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sites selected for the same-day organisation: Patients will be admitted to the hospital and leave it on the same-day of the procedure.
  Interventions: Other: Ambulatory procedure
- Sites with standard overnight hospitalization: Standard organisation with a minimum of one night's stay

INTERVENTIONS:
Other: Ambulatory procedure — In the same-day hospitalization group, some patients will be hospitalized on an ambulatory process
  Groups: Sites selected for the same-day organisation

SUMMARY:
This study has been implemented to evaluate cardiac resynchronization therapy pacemaker (CRT-P) implantations on a same-day basis

DETAILED DESCRIPTION:
The objective of the study is to show in the French centers selected for the same-day organization that a same-day CRT-P implantation is safe, feasible, and associated with significant cost-saving and a minimum conversion rate to full hospitalization by comparing outcomes with patients routinely hospitalized for at least one night. The medical economic evaluation will be based on the SNDS (National Health Data System) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Planned de novo implantation or upgrade to a Cardiac Resynchronization Therapy Pacemaker system according to the intended use
* Patient is able to understand the nature of the registry and has provided written informed consent for BIO|STREAM.HF (heart failure registry) and the registry-based trial BIO|OEDIPE.CRT-P
* Patient enrolled in BIO|STREAM.HF (heart failure registry)

Exclusion Criteria:

* Patients in emergency situation or without medical assessment before hospitalisation for implantation
* Patients previously implanted with an implantable cardiac defibrillator system
* Patients with an implantable cardiac defibrillator indication
* Patients planned to be implanted with an epicardial left ventricular lead (not implanted via the coronary sinus)
* Patients planned to be implanted with His bundle pacing system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients with an indication for a CRT-P system according to current clinical practice and who are already planned to be implanted with a CRT system according to the investigator's decision may be enrolled in this submodule.
Sampling Method: Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events with possible or probable or sure causal relation to the procedure until 6 months after implantation. | over the 6-month follow-up duration
  Number of Serious Adverse Events

SECONDARY OUTCOMES:
Duration of hospitalisation | Time between the patient's entry at the hospital and the patient's hospital discharge, an average of 2 days
  Duration of hospitalisation in days
Evaluation of quality of life | At baseline and 6 months of follow-up
  The patient current health state will be estimated from the answers given by EuroQoL 5D (EQ-5D-5L) questionnaire. The EQ-5D-5L is a self-administered two-part instrument. The first part consists of 5 questions to assess current health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The second part is a 20 centimeters visual analog scale that ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Rate and reason for not selecting patient for a same-day procedure | during the implantation procedure hospitalization
  Number and percentage of patients that were not selected for same-day procedure and the reason why they were not selected for same-day procedure through a questionnaire
Rate and reason for conversion | during the implantation procedure hospitalization
  Number and percentage of patients that were initially elective to same-day procedure but who finally were hospitalized for at least one night and the reason why they were converted to full hospitalization through a questionnaire
Rate of transmitted data by Home Monitoring | through study completion, an average of 6 months
  Number and percentage of data that were transmitted through the Home Monitoring technology
Occurence of atrial and ventricular arrhythmias as detected by Home Monitoring | through study completion, an average of 6 months
  Number of atrial and ventricular arrhythmias as detected by Home Monitoring
Number of persons in charge of analyzing the Home Monitoring data | through study completion, an average of 6 months
  Number of persons in charge of analyzing the Home Monitoring data in each site
Description of the basic programming of the pacemaker | through study completion, an average of 6 months
  Description of the mode that has been chosen by the physician to program the pacemaker
All serious adverse events including patient deaths; all adverse device effects; all cardiovascular adverse events; all device deficiencies | through study completion, an average of 6 months
  Number of each
Chronotropic incompetence and influence of closed loop stimulation on the cardiac resynchronization therapy efficacy | through study completion, an average of 6 months
  Description of the programmation of the chronotropic incompetence
Rate of patients that performed stress tests | through study completion, an average of 6 months
  Number and percentage of patients that performed stress tests
Patient self-assessment | through study completion, an average of 6 months
  Description of the patient self-assessment during follow-ups through a questionnaire : Markedly improved Moderately improved Slightly improved Remained unchanged Slightly worsened Moderately worsened Markedly worsened

OTHER OUTCOMES:
Medico-economic evaluation | through study completion, an average of 6 months
  Cost-utility analysis to compare the efficiency of the same-day and overnight approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Pasquié, Prof., Principal Investigator — University Hospital, Montpellier; Jacques Mansourati, Prof., Principal Investigator — University Hospital, Brest
Locations (19):
- France (19):
  - GCS Centre de Cardiologie du Pays Basque, Bayonne
  - CHU Brest, Brest
  - CHU Caen, Caen
  - Hôpital Louis Pasteur, Chartres
  - Hôpital Saint Philibert, Lomme
  - CH Bretagne Sud, Lorient
  - CHU La Timone, Marseille
  - Hôpital Privé Jacques Cartier, Massy
  - Clinique Les Fontaines, Melun
  - CHU Montpellier, Montpellier
  - Clinique du Millénaire, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Hôpital La Pitié-Salpêtrière, Paris
  - CHU Saint Etienne, Saint-Etienne
  - CH Saint Lô, Saint-Lô
  - Nouvel Hôpital Civil, Strasbourg
  - Clinique Pasteur, Toulouse
  - CHRU de Tours - Hôpital Trousseau, Tours
  - CH Valence, Valence